CLINICAL TRIAL: NCT05825131
Title: A Combination Retrospective and Prospective Natural History Study of Participants With Sanfilippo Syndrome Mucopolysaccharidosis Type IIIC (MPS IIIC)
Brief Title: Natural History Study of Participants With Sanfilippo Syndrome Type IIIC
Acronym: MPSIIIC
Status: Recruiting | Type: Observational
Sponsor: Phoenix Nest (Industry)
Collaborators: Vaincres Les Maladies Lysosomales (Unknown); Association Sanfilippo Sud (Unknown); Aparito Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JLK-447
Record Dates: First submitted 2023-03-23; First posted 2023-04-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Sanfilippo Syndrome Type C
Keywords: Sanfilippo syndrome type C; Mucopolysaccharidosis type III C; MPS IIIC
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood (plasma and serum), cerebrospinal fluid (CSF), urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Retrospective and prospective observational study of patients living with MPS IIIC: Cohort 1: These participants will be a part of the retrospective and prospective Natural History Study, including the C-RARE video assessments. In clinic visits will include: neurocognitive, developmental and behavioral clinical outcome assessments as well as biochemical sample analysis, imaging measures and retrospective medical record review. Participants will record daily living activities through the C-RARE app on their mobile device.
- Remote video recording study and retrospective medical chart review of patients living with MPS IIIC: Cohort 2: These participants will not attend in clinic visits. They will be a part of the C-RARE and retrospective medical chart review analysis. 35 patients with a confirmed diagnosis of MPS IIIC from English, Spanish and Portuguese speaking households will be recruited for this portion of the study.
- Retrospective medical chart review of MPS IIIC patients either living or deceased: Cohort 3: Deceased or living medical record analysis only of patients with MPS IIIC. Living patients will not be participating in cohort 1 clinical study or cohort 2 C-RARE study.

SUMMARY:
This study is planned to document, through retrospective and prospective data collection, syndrome progression in children and young adults with MPS IIIC.

DETAILED DESCRIPTION:
This is a multi-center, natural history study of subjects with Sanfilippo syndrome type C or MPS IIIC. This study will combine a retrospective review of medical records and an ongoing collection of clinical data on an observational basis. Real-world data will be collected at home using a recording device.

Participants will be asked to attend clinic visits in person on a yearly basis. In clinic visits will include neurocognitive, developmental, behavioral, biochemical, imaging measures as well as retrospective medical record analysis.

At 6-month intervals between clinic visits, participants will be contacted remotely for some safety assessments (e.g., collecting information about concomitant medications, concurrent illnesses, and procedure-related adverse events [AEs] and serious AEs [SAEs] since last clinic visit).

At 6-month intervals, caregivers will complete questionnaires and record home video assessments using a dedicated, compliant study application (app) called C-RARE (Recording Application for Real-World Evidence). The C-RARE app consists of 9 tasks of Activities of Daily Living and socialization as well as three parent reported Sanfilippo specific questionnaires.

The objectives of this study are:

* To enhance the understanding of the natural history and progression of MPS IIIC syndrome on behavior, cognitive abilities, mobility, vision, hearing, speech, and expressive and receptive language
* To define and categorize clinical endpoints that may be used in future clinical trials

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of Sanfilippo syndrome type C disease by all of the following:

* Deficiency in heparan-alpha-glucosaminide N-acetyltransferase enzyme activity
* Has presented with signs/symptoms consistent with Sanfilippo syndrome type C, or, for individuals who have not presented with signs/symptoms of disease (eg, siblings of known patients), the determination of eligibility will be at the discretion of the Sponsor in conjunction with the site Investigator
* Genomic DNA analysis demonstrating homozygous or compound heterozygous, pathogenic and/or potentially pathogenic variants in the HGSNAT gene
* Accumulated GAG HS in urine
* Written informed consent from parent or legal guardian and assent from patient, if required
* Parent/legal guardian willing to accompany the patient to all study visits
* Ability to comply with protocol requirements, in the opinion of the Investigator
* Negative urine pregnancy test at screening (nonsterile females of childbearing potential only).

Functional abilities:

* Able to take food or liquid by mouth, able to walk with or without assistance.
* Has an age equivalent on the Vineland Adaptive Behavior Scales (VABS) of ≥1 year.

Exclusion Criteria:

Patients who meet any of the following criteria will not be eligible to participate in the study:

* Have received an investigational drug within 30 days prior to the Baseline Visit
* Concomitant illness or medical condition or extenuating circumstance that, in the opinion of the Investigator, might compromise the patient's ability to comply with protocol requirements, the patient's well-being or safety, or the interpretability of the patient's clinical data
* The presence of significant non-MPS IIIC-related CNS impairment or behavioral disturbances that would confound the scientific rigor or interpretation of results of the study

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a documented diagnosis of Sanfilippo syndrome type C and who are currently untreated with investigational products (drugs/device) for this disease.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Development Quotient (DQ) Using Bayley Scales of Infant Development Assessment Fourth Edition | Baseline, 12 months and 24 months
  The Bayley Scales of Infant and Toddler Development, 4th edition (Bayley-4) is a standardized developmental assessment that provides raw scores for 5 subtests (cognitive, expressive communication, receptive communication, fine motor, gross motor) and standard score norms converted to percentiles for 3 scales (cognition, communication, motor). The Bayley-4 raw scores range from 0-162 for the cognitive subtest, 0-84 for the receptive communication subtest, 0-74 for the expressive communication subtest, 0-92 for the fine motor subtest, and 0-116 for the gross motor subtest; a higher score denotes a better outcome. The Bayley-4 standard score norms are converted to percentiles from <0.1 to >99.9 for the cognitive, language, and motor scales; a higher percentile denotes a better outcome.
Change From Baseline in Vineland Adaptive Behavior Scales Second Edition (VABS-II) Development Quotient (DQ) Score | Baseline, 12 months and 24 months
  The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. The DQ is a means to express a neurodevelopmental/cognitive delay. The DQ was computed as a ratio and expressed as a percentage using the age-equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range, 0, 100). The overall DQ score is calculated from the mean age-equivalent score obtained by averaging out the age-equivalent scores for the all the sub-domains except for Gross and Fine motor skills. This test measures the following 5 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (a composite of the other 4 domains). A positive value indicates improvement in health and cognition.

SECONDARY OUTCOMES:
Change From Baseline on the Color Trail Test Time Score | Baseline, 12 months and 24 months
  Children's Color Trail Test (CCTT) assesses sustained attention, sequencing, and other executive functions while reducing reliance on language. A shorter time to completion denotes a better outcome.
Change From Baseline of Regional Brain Volumes | Baseline, 12 months and 24 months
  Assessed by MRI, and especially cortical grey matter volume (CGMV). The brain MRI will assess volumes of the whole brain, basal ganglia, cerebellum, cerebellar gray matter, cerebellar white matter, cerebral white matter, cortical gray matter, cortical white matter, subcortical gray matter and ventricles; corpus callosum, cortical thickness; and whole brain apparent diffusion coefficient.
Change From Baseline on the Assessment of Behavioral Changes in Sanfilippo (ABCS) | Baseline, 6 months, 12 months, 18 months, 24 months
  There are 12 questions in the ABCS relating to behavior(s) that caregivers of children with Sanfilippo might find challenging to manage. Change from baseline will be determined by raw scores, a higher score denoting improvement in behavior.
Change From Baseline on the Functional Abilities Descriptive Analysis of Type C- Recording Application for Real-world Evidence (C-RARE) | Baseline, 6 months, 12 months, 18 months, 24 months
  Participants functional abilities will be captured via the C- RARE app at baseline, 6 months, 12 months, 18 months, 24 months while performing tasks of Activities of Daily Living (ADLs). ADLs include: Clothing Management, Eating and Drinking, Chewing and Swallowing, Hygiene, Maintaining and Changing positions, Writing Skills, and Walking.
Change From Baseline on the Peabody Picture Vocabulary Test, Fifth Edition | Baseline, 12 months, 24 months
  The PPVT-5 is a norm-referenced and individually administered measure of receptive vocabulary. Upon hearing a word, the child will be asked to indicate (by pointing) which picture among four options is specified.
Change From Baseline on the Expressive Vocabulary Test Third Edition | Baseline, 12 months, 24 months
  The EVT-3 is a norm-referenced and individually administered test of expressive language.
Change From Baseline in Speech Through Picture Description | Baseline, 12 months, 24 months
  Picture Description will be used to measure speech rate, utterance length, grammatical competence, lexical retrieval ability, and motor speech features in subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Guffon, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States
- Hospices Civils De Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided
The data collected as part of the observational study may be analyzed and published. Phoenix Nest recognizes the importance of communicating medical study data and therefore encourages the publication of these data in reputable scientific journals and at seminars or conferences. The details of the processes of producing and reviewing reports, manuscripts, and presentations based on the data from this study will be described in the Clinical Trial Agreement between Phoenix Nest and the Investigator/institution. Consideration for authorship of all publications will be based on compliance with the Uniform Requirements for Manuscripts Submitted to Biomedical Journals ("Uniform Requirements") of the International Committee of Medical Journal Editors (http://www.icmje.org/ethical_1author.html) and Good Publication Practices.